CLINICAL TRIAL: NCT04684862
Title: Combined Infusion System to Deliver Chemotherapy Regionally to the Liver
Brief Title: Infusion System for Hepatic Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ronald DeMatteo, M.D. (Other)
Responsible Party: Sponsor-Investigator, Ronald DeMatteo, M.D., Chair, Department of Surgery; John Rhea Barton Professor of Surgery, Abramson Cancer Center at Penn Medicine
Organization: Abramson Cancer Center at Penn Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 19220
Record Dates: First submitted 2020-12-22; First posted 2020-12-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer Metastatic to Liver; Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Hepatic Artery Infusion (HAI) Therapy (Experimental): Eligible patients will be implanted with a device that combines components of two commercially available drug delivery pumps to administer regional chemotherapy (FUDR) to the liver. Specifically, a Medtronic pump is being used with an Intera tapered catheter, instead of the Medtronic catheter.
  Interventions: Device: Medtronic SynchroMed II programmable pump connected to an Intera tapered catheter (Combined Infusion System)

INTERVENTIONS:
Device: Medtronic SynchroMed II programmable pump connected to an Intera tapered catheter (Combined Infusion System) — This infusion system is composed of a Medtronic SynchroMed II programmable pump connected to a Intera tapered catheter. Specifically, the Medtronic pump comes with a small connector that ends in a metal flange. During the operation, under sterile conditions, the distal 1 cm of the flange is severed using a scissor. Then, using a Intera connector pin, the end of the Medtronic catheter is connected to the Intera catheter . Two 2-0 silk ties secure the catheters to the pin. The pump and catheter are then inserted into the patient into the abdominal wall or into the chest wall. The catheter is inserted into an artery within the abdomen (usually the gastroduodenal artery but it depends on the exact arterial branching in the individual patient) that feeds the liver.

SUMMARY:
This is a single-site, open-label continued access study/treatment protocol under a treatment IDE. In addition to treating patients, the primary objective of this study is to assess the safety of using the Medtronic SynchroMed II programmable pump combined with the Intera tapered catheter for hepatic artery infusion (HAI) of a standard chemotherapy (FUDR) drug for adults with a clinical or biopsy-proven diagnosis of colorectal cancer metastatic to the liver or intrahepatic cholangiocarcinoma.

After successful implantation, the combined pump and catheter system will be evaluated using a nuclear scan in the postoperative period, which is standard procedure to confirm that the pump is functioning prior to HAI of FUDR. Monitoring for safety will include a record of residual pump volume when it is emptied (every 2-12 weeks depending on whether the pump is being used for chemotherapy infusion) to determine if the pump is still working and surveillance of routine cross-sectional imaging (usually every 2-6 months) for any sign of a pump or catheter problem. Patients will be monitored for the safety of the pump/catheter combination for up to 5 years or pump removal/study withdrawal.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be greater than or equal to 18 years of age
* Have a clinical or biopsy-proven diagnosis of colorectal cancer metastatic to liver or intrahepatic cholangiocarcinoma
* At the time of pump placement, patients will either have unresectable, chemotherapy-responsive disease or they will be undergoing resection with planned postoperative HAI
* Be deemed appropriate for pump chemotherapy by both a medical oncologist and a surgical oncologist
* Provision of signed and dated informed consent form

Exclusion Criteria:

* Known active infection
* Is pregnant or breastfeeding or expecting to conceive children within the projected duration of the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-08 (Actual); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Number of Targeted Adverse Events (TAEs) | From surgery up to 60 months post-surgery or study withdrawal
  TAEs are defined as AEs deemed related to the combination of the devices (i.e., the connection between the Medtronic pump and Intera Catheter).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States